CLINICAL TRIAL: NCT06276062
Title: Short Term Functional and Radiological Outcomes of Using Double Short Titanium Elastic Nails in Treatment of Pediatric Distal Radius Fractures.
Brief Title: Uses of Titanium Nail in Pediatric Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Abdellah Desoky, Principal Investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Titanium nail usage
Record Dates: First submitted 2024-02-18; First posted 2024-02-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Trauma Injury of Upper Extremity Forearm Multiple; Fracture of Distal End of Radius
Keywords: Pediatric Trauma; fractures; Double Titanium nail; Distal Radial Fractures; Intramedullary nail fixation
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pediatric distal radial fractures. (Experimental): Pediatric traumatized patients aged between 4 to 16 years old who presented by distal radial fractures and need to go under operative management.
  Interventions: Procedure: Distal radius fracture fixation in pediatrics.

INTERVENTIONS:
Procedure: Distal radius fracture fixation in pediatrics. — using double short titanium elastic nails in treatment of pediatric distal radius fractures.

SUMMARY:
The aim of this study is to investigate the short term functional and radiological outcomes of using double short titanium elastic nails as treatment of pediatric distal radius fractures.

DETAILED DESCRIPTION:
Severely displaced distal radial fractures in children are generally considered unstable; especially when associated with total rupture of the periosteum. Although the remodeling potential of distal radial fractures is very good in childhood, a subgroup of severely displaced and unstable distal pediatric forearm fractures are candidates for operative fixation because acceptable reduction cannot be maintained in a conservative way. These injuries are usually candidates for closed reduction and minimal invasive fixation.

Operative osteosynthesis technique of pediatric wrist fractures are optimally minimally invasive, physeal sparing, and with acceptable reduction.

Most operative methods need complementary 4 to 6 weeks of postoperative immobilization by casting. Many of these techniques do not respect physeal plates. Both current available fixation techniques; modifications of Kirschner wiring or conventional elastic stable intramedullary nailing [ESIN]) have the same rate of mild complications. Growth disturbance is a rare, but represents a very rare severe complication of transepiphyseal wire placement.

Varga et al. Medicine (2017) 96:14[8] used modified ESIN method for operative treatment of severely displaced pediatric distal metaphyseal or metadiaphyseal radial fractures. With 2 short, prebent, retrograde elastic titanium nails inserted proximal to the distal radial physis, a very stable stabilization achieved without the need for a prolonged period of cast immobilization. The nails do not cross the physeal plates, so the possibility of postoperative physeal arrest is reduced.

their results:(the study shows a new technique in fixation of severely displaced pediatric distal radial fractures é more stable fixation,less pin track irritations and infections,early return to full range of motion within the sixth postoperative week, short removable splint was sufﬁcient for early pain-free mobilization.

All the x-rays made 6 months postoperatively showed anatomic reduction, and there has been no sign of omic reduction, and there has been no sign of growth disturbance at the area of thece at the area of the distal radius) We conduct this study to evaluate the Short term functional and radiological outcomes of using double short titanium elastic nails in treatment of pediatric distal radius fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patient Age ( 4 - 16 ) Years old.
* Both sex included .
* Simple or compound fractures (Grade I).
* Isolated fracture in the limb.
* Severely displaced fracture (Angulated).
* Recent and old distal radius fractures

Exclusion Criteria:

* Ages below 4 years or above 16 years.
* Associated with other fractures in the same limb.
* Compound fractures ( Grade II,III).
* Comminuted or Pathological fractures.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Comparison between usage of titanium nail and old methods | 2 Weeks up to 6 Weeks
  As old techniques used to reduce severely displaced fracture, the new technique assures better healing and full range motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varga M, Jozsa G, Fadgyas B, Kassai T, Renner A. Short, double elastic nailing of severely displaced distal pediatric radial fractures: A new method for stable fixation. Medicine (Baltimore). 2017 Apr;96(14):e6532. doi: 10.1097/MD.0000000000006532. PMID 28383417